CLINICAL TRIAL: NCT06667024
Title: Dexmedetomidine as an Intrathecal Adjuvant to Hyperbaric Bupivacaine for Postoperative Analgesia in Patients Undergoing Arthroscopic Anterior Cruciate Ligament Reconstruction Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Abdallah Elsayed Elkasrawy, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS288/8/23
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Dexmedetomidine; Intrathecal; Adjuvant; Hyperbaric Bupivacaine; Analgesia; Arthroscopic Anterior Cruciate Ligament Reconstruction
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients received the standard spinal anesthesia with 0.5% 3 ml according to the patient hyperbaric bupivacaine only.
  Interventions: Drug: Hyperbaric bupivacaine
- Dexmedetomidine (study) group (Experimental): Patients received dexmedetomidine 4 μg and 0.5% (3-4 ml according to the patient's height) hyperbaric bupivacaine.
  Interventions: Drug: Dexmedetomidine and Hyperbaric bupivacaine

INTERVENTIONS:
Drug: Hyperbaric bupivacaine — Patients received the standard spinal anesthesia with 0.5% 3 ml according to the patient hyperbaric bupivacaine only
  Arms: Control group
Drug: Dexmedetomidine and Hyperbaric bupivacaine — Patients received dexmedetomidine 4 μg and 0.5% (3-4 ml according to the patient height) hyperbaric bupivacaine
  Arms: Dexmedetomidine (study) group

SUMMARY:
This study aimed to evaluate the effect of adding low doses of dexmedetomidine to hyperbaric bupivacaine during spinal anesthesia on post operative analgesia characteristics in Arthroscopic Anterior Cruciate Ligament Reconstruction Surgeries

DETAILED DESCRIPTION:
The anterior cruciate ligament (ACL) is injured frequently during sports participation. Arthroscopic evaluation of patients with acute traumatic hemarthrosis of the knee has repeatedly demonstrated a 60% to 70% incidence of ACL injury.

Postoperative pain should be effectively treated because it represents an important component of postoperative recovery. Effective treatment serves to blunt autonomic, somatic, and endocrine reflexes with a resultant potential decrease in perioperative morbidity.

Dexmedetomidine is a highly selective α2-adrenergic agonist that has been used for premedication and as an adjunct to general anesthesia. It reduces opioid and inhalational anesthetics requirements.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 21 to 50 years.
* Both genders.
* American society of anesthesiologists (ASA) physical status I and II.
* Patients scheduled for arthroscopic anterior cruciate ligament reconstruction surgeries under spinal anesthesia.

Exclusion Criteria:

* Patient refusal.
* Body Mass Index (BMI) more than 40 kg/m2.
* Patients who were taking analgesics for chronic pain on opioid therapy or have a history of drug abuse.
* Uncooperative patient.
* Patients with coagulation disorders.
* History of local anesthetics allergy.
* Infection at the needle puncture site.
* Patients with significant respiratory, cardiac, renal or hepatic disorders

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  The rescue analgesia was morphine IV bolus of 3 mg with when VAS > 30. Total morphine consumption in the first 24 hours postoperatively was documented.

SECONDARY OUTCOMES:
Time to first rescue analgesia request | 24 hours postoperatively
  Time to the first rescue analgesia (time from end of surgery to first dose of morphine administrated) was recorded
Degree of pain | 24 hours postoperatively
  Degree of pain was assessed using Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 100 represents "the worst pain imaginable"). VAS was assessed at PACU, 1, 2, 4, 8, 12, 18, 24 hours postoperatively.
Duration of motor block | Intraoperatively
  Duration of motor block starting from the time when the Bromage score 3 after spinal anesthesia until the time when the Bromage score was 0 postoperative.
Patient satisfaction | 24 hours postoperatively
  Patients' satisfaction was measured 24 hours postoperative using a five-point Likert scale consisting of:
  1: Very dissatisfied, 2: Dissatisfied, 3: Unsure, 4: Satisfied, 5: Very satisfied
Incidence of side effects | 24 hours postoperatively
  Incidence of side effects such as Hypotension, Bradycardia, Shivering, nausea, and vomiting) were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.